CLINICAL TRIAL: NCT03430297
Title: A Randomized, Controlled, Multi-center, Phase III Clinical Study to Investigate Recombinant Humanized PD-1 Monoclonal Antibody Injection (JS001) Versus Dacarbazine as the 1st-line Therapy for Unresectable or Metastatic Melanoma
Acronym: JS001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMO-JS001-III-MM-01
Record Dates: First submitted 2018-01-29; First posted 2018-02-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Melanoma; Unresectable Melanoma
Keywords: anti-PD-1 monoclonal antibody; the First Line Therapy; Dacarbazine; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 240mg Q2W (Experimental)
  Interventions: Biological: JS001 240mg Q2W
- Dacarbazine 1000mg/m2 Q3W (Active Comparator)
  Interventions: Drug: Dacarbazine 1000mg/m2 Q3W

INTERVENTIONS:
Biological: JS001 240mg Q2W — recombinant humanized anti-PD-1 monoclonal antibody injection (JS001) will be provided by the sponsor. Strength: 240mg/6ml/vial. 240mg, once every two weeks.
  Control drug: dacarbazine (1000mg/m2, d1, intravenously, once every three weeks). The dose will be given intravenously over 180 minutes (the infusion time can be prolonged according to the institutional criteria), starting from Week 1, once every 3 weeks, until progression of disease.
  Arms: JS001 240mg Q2W
Drug: Dacarbazine 1000mg/m2 Q3W — The dose of DTIC will be calculated according to the following formula, where the 'X' represents the total mg dose of DTIC: X (mg) = [body surface area (BSA) x (1000mg/m2)].
  The body surface area (BSA) is defined by Dubois formula: BSA (m2) = 0.007184* (cm0.725) * (kg0.425)
  Arms: Dacarbazine 1000mg/m2 Q3W

SUMMARY:
This is one phase III, randomized, open-label study in comparison of JS001 with dacarbazine as the 1st-line therapy for adult (≥18 years) subjects with unresectable or metastatic melanoma. The subjects will be 1:1 randomized and stratified in accordance with acral lentiginous melanoma and M stage (M0vsM1a/M1bvsM1c). Using standard dose and dose interval, the subjects will be given JS001 240mg intravenously, once every two weeks, or dacarbazine 1000mg/m2, d1, intravenously, once every three weeks. One cycle of therapy is 6 weeks (3 doses of JS001 or 2 doses of dacarbazine per cycle).

DETAILED DESCRIPTION:
1. In the subjects who have clinical benefit evaluated by investigators and tolerate the study treatment, treatment will be considered to give after occurrence of progression defined by RECIST1.1 as evaluated by the initial investigators, these subjects must terminate the treatment when further progression is validated.
2. The subjects in dacarbazine treatment group are allowed to be crossed to receive JS001 after progression of disease; however, they need to be re-evaluated if they meet the inclusion/exclusion criteria.

Subjects need to provide one tumor tissue specimen for archival or one newly acquired biopsy tissue from the site that is previously not irradiated for evaluation of PD-L1 expression status when they participate in the study. The PD-L1 expression status of specimen will be evaluated in the central laboratory using immunohistochemical (IHC) method. Subjects with positive or negative PD-L1 can be enrolled in this study, and the clinical activity in the two subgroups will be evaluated in accordance with the prespecified subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for participation in the trial only when they meet the following criteria:
* Age ≥18 years, male or female;
* Systemic treatment-naïve, histologically confirmed unresectable stage III or IV melanoma. Previous adjuvant or neoadjuvant therapy is allowed, however, it is required to be completed at least three weeks prior to the randomization, and all the relevant adverse events have been recovered to normal or CTC-AE grade 1;
* Measurable lesion (according to RECIST v1.1 criteria);
* ECOG score 0 or 1
* Tumor tissue has to be provided (FFPE archival or newly acquired tissue block or unstained slide from FFPE) for analysis of biomarkers;
* Previous radiotherapy must be completed at least two weeks prior to administration of investigational product;
* The laboratory data for screening must meet the following criteria and should be acquired within 14 days prior to the first dose:

  1. Peripheral hemogram: white blood cell (WBC) ≥3.0×109/L, neutrophil (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (Hgb) ≥90g/L;
  2. Renal function: serum creatinine°≤1.5 x ULN or calculated creatinine clearance (CrCl) >40 mL/min (using Cockcroft Gault formula);
  3. Hepatic function: AST/ALT≤2.5 x ULN in subjects without hepatic metastasis, AST/ALT≤5 x ULN in those with hepatic metastasis;
  4. Total bilirubin ≤1.5 x ULN (except the subjects with Gilbert syndrome, the total bilirubin must be < 3.0mg/dL).
* Estimated survival ≥16 weeks;
* Men with reproductive capacity or women of childbearing potential must use highly effective contraceptive methods during the trial (e.g., oral contraceptives, intrauterine device, sexual abstinence or barrier method combined with spermicide), and continue contraception for 12 months after the end of treatment;
* Subject is willing to participate in the study, sign the informed consent form with good compliance and cooperation with follow-up;
* Re-enrollment: re-enrollment of subjects who discontinue the study for failure prior to the treatment (i.e., the subject has not been randomized/received any treatment yet) is allowed in this study. The subjects must re-sign the informed consent form if they are re-enrolled.

Exclusion Criteria:

* Patients will be excluded from the trial when they have any one of the following conditions:
* Previous treatment with anti-PD-1, anti-PD-L1or anti-PD-L2 therapy;
* Known allergy to recombinant humanized anti-PD-1 monoclonal antibody and its components;
* Presence of BRAF mutation, except unwillingness or inability to receive BRAF mutation inhibitor;
* Malignant melanoma originated from eyes or mucosa;
* Having received other anti-tumor therapy (including corticosteroids, immunotherapy) or participated in other clinical studies within 4 weeks prior to the start of treatment, or having not recovered from the previous toxicity (except grade 2 alopecia and grade 1 neurotoxicity);
* Pregnant or lactating women;
* HIV positive; HCV positive; positive HBV DNA copies detected simultaneously with HBsAg or HBCAb positive (quantitative detection limit 500 IU/ml);
* History of active pulmonary tuberculosis;
* Active autoimmune disease requiring systemic treatment in the past two years (e.g., use of disease-modulating drugs, corticosteroids or immunosuppressive drugs), relevant alternative therapy is allowed (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency);
* Other serious, uncontrollable concomitant diseases that may affect the compliance with protocol or interfere with interpretation of the results, including active opportunistic infection (serious) infection in progressive stage, uncontrollable diabetes, cardiovascular disease (grade Ⅲ or Ⅳ heart failure defined by New York Heart Association, degree Ⅱ and above cardiac block, myocardial infarction in the past 6 months, unstable arrhythmia or unstable angina pectoris, cerebral infarction within 3 months, etc.) or pulmonary disease (history of interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm);
* Subjects with active central nervous system (CNS) metastasis, active brain metastasis or leptomeningeal metastatic foci. For the subjects with brain metastasis, if they have received treatment and have no evidence of progressive disease on the nuclear magnetic resonance imaging (MRI) at least 8 weeks after completion of the treatment and within 28 days prior to the first dose, they are eligible to participate in the study. Meanwhile, it is required corticosteroid for systemic therapy at the dose of immunosuppressant (>10mg/day prednisone equivalent) must not be needed at least two weeks prior to administration of investigational product;
* Previously receiving hematopoietic stimulating factor within two weeks prior to the start of treatment, for example, colony stimulating factor, erythropoietin;
* Having been injected by live vaccine within 4 weeks prior to the start of treatment;
* Major surgery within 4 weeks prior to the start of treatment (not including diagnostic surgery);
* History of psychotropic drug abuse and inability to give up or history of mental disorder;
* Having other malignant tumors that have not been recovered in the past 5 years, not including obviously cured malignancies, or curable cancers, for example, basal cell carcinoma or squamous cell cutaneous carcinoma, superficial bladder cancer or carcinoma in situ of prostate, carcinoma in situ of cervix or carcinoma in situ of breast;
* Other severe, acute or chronic medical or mental diseases or abnormal laboratory findings that may increase the risk from participation in the study, or interfere with interpretation of study results according to investigators' opinion.

Eligibility criteria on cross-over to JS001 treatment period -inclusion criteria for the subjects who are previously randomized into DTIC:

* According to investigators' evaluation, the subjects must have documented radiological progression of disease during DTIC treatment;
* Previous anticancer therapy, including DTIC and palliative radiotherapy, must be completed at least three weeks prior to the dose of JS001;
* Adverse events related with DTIC or palliative radiotherapy must have been relieved to grade 1 or baseline at randomization;
* Any major surgery must be completed at least 28 days prior to the first dose of JS001;
* No previous treatment with anti-PD-1 or anti-PD-L1 therapy;
* The laboratory data on the eligibility for cross-over therapy must meet the following criteria and should be acquired within 14 days prior to the start of JS001 treatment:
* Peripheral hemogram: white blood cell (WBC) ≥3.0×109/L, neutrophil (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (Hgb) ≥90g/L;
* Renal function: serum creatinine≤1.5 x ULN or calculated creatinine clearance (CrCl) >40 mL/min (using Cockcroft Gault formula);
* Hepatic function: AST/ALT≤2.5 x ULN in subjects with no hepatic metastasis, AST/ALT≤5 x ULN in those with hepatic metastasis;
* Total bilirubin≤1.5 x ULN (except the subjects with Gilbert syndrome, total bilirubin must be<3.0mg/dL).
* Men with reproductive capacity or women of childbearing potential must use highly effective contraceptive methods during the trial (e.g., oral contraceptives, intrauterine device, sexual abstinence or barrier method combined with spermicide), and continue contraception for 12 months after the end of treatment;
* Subjects are willing to participate in the study, sign the informed consent form with good compliance and cooperation with follow-up;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
the progression-free survival (PFS) | 3 months
  To compare the progression-free survival (PFS) evaluated by one independent review board of radiological data in systemic treatment-naïve patients with unresectable, locally advanced or metastatic melanoma who are treated with JS001 versus dacarbazine.

SECONDARY OUTCOMES:
objective response rate (ORR) | 2 years
  To compare objective response rate (ORR) evaluated by the independent review board of radiological data according to RECIST 1.1 between the two groups;
duration of response (DOR) | 2 years
  To compare duration of response (DOR) evaluated by the independent review board of radiological data according to RECIST 1.1 between the two groups;
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (11):
- China (11):
  - Hefei Binhu Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital Of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng X, Huang G, Fang M, Li K, Wu D, Zhang X, Chen J, Zhu D, Chen Y, Li H, Gao Q, Wu L, Tang B, Yan X, Zeng R, Li J, Yu W, Xu J, Hao Y, Jin C, Zou J, Guo J. Toripalimab vs Dacarbazine as First-Line Therapy for Advanced Melanoma of Acral Subtype: The Phase 3 MELATORCH Randomized Clinical Trial. JAMA Oncol. 2026 Jan 2:e255751. doi: 10.1001/jamaoncol.2025.5751. Online ahead of print. PMID 41481311